CLINICAL TRIAL: NCT02387476
Title: Non-Inferiority Study of the FRESCA Mask Versus Existing CPAP Mask for Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FRESCA Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000-01
Record Dates: First submitted 2014-10-14; First posted 2015-03-13 (Estimated); Results first posted 2018-03-23 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea; OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FRESCA mask first night (Experimental): FRESCA mask first night (experimental device) | CPAP second night (active comparator)
  Interventions: Device: FRESCA mask first night; Device: CPAP Mask first night
- CPAP Mask first night (Experimental): CPAP Mask first night (active comparator)| FRESCA mask second night (experimental device)
  Interventions: Device: FRESCA mask first night; Device: CPAP Mask first night

INTERVENTIONS:
Device: FRESCA mask first night — FRESCA nasal mask first night
Device: CPAP Mask first night — CPAP Nasal Mask first night

SUMMARY:
This will be a prospective study in subjects with Obstructive Sleep Apnea (OSA) to characterize the clinical performance during a single night of therapy with a FRESCA mask compared with a single night of therapy with their existing nasal Continuous Positive Airway Pressure (CPAP) mask.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a common chronic disorder and the most common of all sleep disorders. OSA can occur in any age group, but prevalence increases between middle and older age. Over the last two decades the prevalence of sleep disordered breathing seems to be increasing in both men and women, likely due to increasing rates of obesity. Relative increases reported are between 14% and 55% depending on the subgroup. For men, the current prevalence estimates of moderate to severe sleep-disordered breathing are 10% for 30 to 49 year-olds and 17% for 50 to 70 year-olds. For women, the corresponding prevalence estimates are 3% and 9%.

Common consequences of OSA include daytime sleepiness, extreme daytime fatigue, slow reaction time, moodiness, belligerence and vision problems. OSA is also linked to hypertension, increased cardiovascular morbidity, type 2 diabetes, neurocognitive dysfunction and possibly cancer.

The study is a prospective, comparative, open label, randomized crossover assignment, multi-center pivotal study.

Up to forty-five (45) subjects will be enrolled. It is desirable to have the subject population distributed across the OSA severity criteria range.

The purpose of this study is to demonstrate that the FRESCA mask is non-inferior to a CPAP nasal mask in maintaining AHI and ODI during a single night of PSG assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 18-70 years old;
2. Qualifying diagnostic polysomnography (PSG): Resulting in AHI > 5/hr of sleep (using conventional lab or home test);
3. Qualifying titration PSG: In lab titration within the past 12 months and therapeutic pressure resulting in Apnea Hypopnea Index (AHI) < 5/hr;
4. Primary medical diagnosis of OSA/ Hypopnea syndrome and on CPAP treatment > 1 month;
5. Current user of nasal mask or nasal pillow mask;
6. Have regular usage of their CPAP machine ( at least 4 hrs per night and at least 5 nights per week) confirmed by secure digital (SD) card download;
7. No significant changes in the subject's general health and no change in weight greater than ±10 lbs since titration PSG was performed and CPAP therapy initiated (confirmed from medical records);
8. BMI < 35 kg/m2;
9. Must be able to be fit properly with FRESCA mask;
10. Must be able to comply with all study requirements as outlined in the protocol;
11. Must be able to understand English and be willing to provide written informed consent.

Exclusion Criteria:

1. Subjects with non OSA sleep disorders;
2. Substantial central or mixed apneas (Central and Mixed apnea index ≥ 5/hr);
3. Subjects actively using bi-level PAP or require oxygen therapy;
4. Subjects using a full face mask or chin strap;
5. History of severe cardiovascular disease, including New York Heart Association (NYHA) Class III or IV heart failure, coronary artery disease (CAD) with angina or myocardial infarction (MI)/stroke within past 6 months;
6. Subjects who are medically complicated or who are medically unstable (i.e. cancer, dementia, unstable cardiac or respiratory disease, or unstable psychiatric illness);
7. Potential sleep apnea complications that in the opinion of the investigator may affect the health and safety of the participant including: uncontrolled hypertension or hypotension, low blood oxygen (oxygen desaturations nadirs below 75% on their diagnostic PSG), or use of medication or other treatment which may pose additional risk to the subject;
8. Subjects exhibiting any flu-like or any upper airway tract infection symptoms at time of assessment;
9. Subjects with ongoing severe nasal allergies or sinusitis or difficulty breathing through the nose; persistent blockage or one or both nostrils; or any nasal or facial abnormalities that would not allow adequate placement of the device;
10. Subjects with prior surgical intervention for obstructive sleep hypopnea/ apnea syndrome;
11. Currently working nights, rotating night shifts, planned travel across two or more time zones required during study period, or within two weeks prior to study enrollment, or sleep schedule not compatible with sleep lab practices;
12. Unstable use of medications or other agents that may affect sleep or PSG (sedatives or hypnotics);
13. Pregnant (confirmed verbally);
14. Consumption of > 500mg caffeine per day (e.g. > 8 cola-type beverages, > 5 cups of coffee);
15. Currently enrolled in any other research study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — FRESCA Medical
Locations (5):
- United States (5):
  - Sequoia Sleep Diagnostics, Fresno, California
  - Complete Sleep Solutions, Murrieta, California
  - Broward Research Group, Hollywood, Florida
  - CliniLabs, Inc, New York, New York
  - SleepMed of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven (11) subjects were not included in the primary analysis due to incomplete data on at least one PSG nights.
  mITT Group (subjects completing 2 nights on study with a Valid PSG result) n=36 See section 8.1 of Clinical Study Report (TR 1000-01) for details.
Groups:
- FRESCA Mask First - CPAP Second: First night using FRESCA nasal mask and second night using CPAP
  FRESCA Nasal Mask: FRESCA nasal mask
- CPAP Mask - FRESCA Mask Second: One night using CPAP nasal mask and then second night using FRESCA nasal mask
  CPAP Nasal Mask: CPAP nasal pillow and nasal mask
Period: Overall Study
Arm/Group | FRESCA Mask First - CPAP Second | CPAP Mask - FRESCA Mask Second
Started | 25 | 22
Completed | 19 | 17
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- FRESCA Mask First CPAP Mask Second: One night using FRESCA nasal mask and the second night using patient provided CPAP
- CPAP Mask First and CPAP Mask Second: One night using patient providing CPAP nasal mask and second night using FRESCA mask
- Total: Total of all reporting groups
Arm/Group | FRESCA Mask First CPAP Mask Second | CPAP Mask First and CPAP Mask Second | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Customized [Count of Participants; unit: Participants]
  Age: age less than 18 years old | 0 | 0 | 0
  Age: age between 18-70 years old | 19 | 17 | 36
  Age: age less than 70 years old | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 13 | 13 | 26
Apnea-Hypopnea Index >= 5/hr [Mean (Standard Deviation); unit: events/hour] | 23.6 (15.317) | 28.8 (19.571) | 26.1 (17.403)
BMI<= 35 kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 30.91 (2.961) | 29.89 (3.543) | 30.43 (3.242)

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: The Apnea-Hypopnea Index or Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. Difference of AHI values between patients who used the FRESCA treatment first versus the CPAP treatment.
Time Frame: per hour
Population: The population for analysis for the primary outcomes is the modified Intent-to-Treat (mITT) population. This population consists of the enrolled, intent-to-treat population who has evaluable data for both nights of PSG evaluation.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- FRESCA Mask First Night: First night using FRESCA nasal mask and second night using CPAP
  FRESCA Nasal Mask: FRESCA nasal mask
- CPAP Mask First Night: One night using CPAP nasal mask and then second night using FRESCA nasal mask
  CPAP Nasal Mask: CPAP nasal pillow and nasal mask
Arm/Group | FRESCA Mask First Night | CPAP Mask First Night
Number analyzed (Participants) | 19 | 17
events per hour
  First Night | 1.96 (3.414) | 3.73 (8.565)
  Second Night | 1.23 (1.526) | 4.12 (5.857)
  Overall | 2.98 (4.783) | 2.41 (6.028)
Statistical Analysis 1: Comparison: FRESCA Mask First Night vs CPAP Mask First Night; This analysis was planned to assume a non-inferiority (NI) margin of 5 units and a 1-sided alpha level of 2.5%. A 2-sided 95% confidence interval (CI) was also planned to be provided around the difference between treatments, where non-inferiority would also be demonstrated if the upper bound of the 95% CI is less than or equal to the NI margin of 5 units. In this scenario, the 2-sided 95% CI equates to testing the 1-sided non-inferiority hypothesis; Test type: Non-Inferiority — This analysis was planned to assume a non-inferiority (NI) margin of 5 units and a 1-sided alpha level of 2.5%. A 2-sided 95% confidence interval (CI) was also planned to be provided around the difference between treatments, where non-inferiority would also be demonstrated if the upper bound of the 95% CI is less than or equal to the NI margin of 5 units. In this scenario, the 2-sided 95% CI equates to testing the 1-sided non-inferiority hypothesis; p < 0.001, t-test, 1 sided — The p-value to test non-inferiority of FRESCA Mask compared with CPAP Mask (FRESCA-CPAP<5 units) assumes a 1-sided test using a level of significance of 2.5% and NI margin of 5 units; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.7 to 2.9], Standard Deviation 1.13 — The mean AHI is rounded to a single decimal point in the text of the report (3.0 and 2.4, respectively), in order to be consistent with standard reporting of AHI

2. Primary Outcome: Oxygen Desaturation Index (ODI)
Description: The Oxygen Desaturation Index (ODI) is the number of times per hour of sleep that the blood's oxygen level drop by a certain degree from baseline. The ODI is typically measured as part of standard sleep studies, such as a diagnostic polysomnogram, home sleep apnea testing, or with overnight oximetry.Difference of ODI values between patients who used the FRESCA treatment first versus the CPAP treatment.
Time Frame: per hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | FRESCA Mask First Night | CPAP Mask First Night
Number analyzed (Participants) | 19 | 17
events per hour
  First Night | 1.11 (1.730) | 1.2 (2.530)
  Second Night | 1.05 (1.569) | 1.7 (2.364)
  Overall | 1.39 (2.046) | 1.12 (2.049)
Statistical Analysis 1: Comparison: FRESCA Mask First Night vs CPAP Mask First Night; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.4 to 1.0], Standard Deviation 0.36 — The mean ODI values are rounded to a single decimal point value in the text of the table (1.4 and 1.1, respectively) to ensure consistency with ODI reporting standards

3. Secondary Outcome: Arousal Index (AI)
Description: The number of arousals per hour; arousals are defined as a change in EEG for at least 3 seconds.
Time Frame: per hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | FRESCA Mask First Night | CPAP Mask First Night
Number analyzed (Participants) | 19 | 17
events per hour
  First Night | 21.95 (15.572) | 20.94 (8.728)
  Second Night | 17.32 (8.083) | 24.00 (8.895)
  Overall | 22.92 (12.727) | 19.03 (8.473)

4. Secondary Outcome: Sleep Efficiency (SE%)
Description: Sleep Efficiency (%) [100 x Total sleep time/ total recording time] reported per treatment
Time Frame: per night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency
Groups:
- FRESCA Mask First Night | CPAP Second Night: First night using FRESCA nasal mask and second night using CPAP
  FRESCA Nasal Mask: FRESCA nasal mask
- CPAP Mask First Night | FRESCA Mask Second Night: One night using CPAP nasal mask and then second night using FRESCA nasal mask
  CPAP Nasal Mask: CPAP nasal pillow and nasal mask
Arm/Group | FRESCA Mask First Night | CPAP Second Night | CPAP Mask First Night | FRESCA Mask Second Night
Number analyzed (Participants) | 19 | 17
percentage of sleep efficiency
  First Night | 80.63 (7.697) | 84.47 (11.549)
  Second Night | 86.68 (7.212) | 78 (9.192)
  Overall | 79.39 (8.419) | 85.64 (9.433)

5. Secondary Outcome: Minimum Sleep SpO2 (%)
Description: The minimum O2 level percentage during treatment reported per treatment
Time Frame: per night
Measure: Mean (Standard Deviation); unit: percentage of O2 Saturation
Arm/Group | FRESCA Mask First Night | CPAP Second Night | CPAP Mask First Night | FRESCA Mask Second Night
Number analyzed (Participants) | 19 | 17
percentage of O2 Saturation
  First Night | 89.16 (3.775) | 91.41 (3.858)
  Second Night | 91.95 (2.321) | 89.06 (5.517)
  Overall | 89.11 (4.609) | 91.69 (3.106)

6. Secondary Outcome: Mean Sleep SpO2 -(%)
Description: Mean Sleep SpO2 - blood oxygenation level (%) mean value reported per treatment
Time Frame: per night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of O2 Saturation
Arm/Group | FRESCA Mask First Night | CPAP Second Night | CPAP Mask First Night | FRESCA Mask Second Night
Number analyzed (Participants) | 19 | 17
percentage of O2 Saturation
  First Night | 94.89 (1.41) | 95.35 (1.498)
  Second Night | 95 (1.414) | 95.41 (1.326)
  Overall | 95.14 (1.376) | 95.17 (1.444)

7. Secondary Outcome: Wakefulness (Min)
Description: Measure of time not sleeping (minutes)
Time Frame: per night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FRESCA Mask First Night | CPAP Mask First Night
Number analyzed (Participants) | 19 | 17
minutes
  First Night | 78.95 (35.68) | 61.06 (58.463)
  Second Night | 51.79 (32.898) | 90.88 (44.933)
  Overall | 84.58 (40.177) | 56.17 (45.272)

8. Secondary Outcome: Stage N1 (Min)
Description: Stage N1 sleep is an estimate of the degree of sleep fragmentation.
Time Frame: per night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FRESCA Mask First Night | CPAP Second Night | CPAP Mask First Night | FRESCA Mask Second Night
Number analyzed (Participants) | 19 | 17
minutes
  First Night | 43.53 (20.614) | 49.88 (19.906)
  Second Night | 40.26 (18.363) | 53.47 (25.873)

9. Secondary Outcome: Stage N2 (Min)
Description: Stage N2 sleep predominates the sleep stages with 50% of the total sleep time. It follows the Stage N1 sleep and continues to recur throughout the night.
Time Frame: per night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FRESCA Mask First Night | CPAP Second Night | CPAP Mask First Night | FRESCA Mask Second Night
Number analyzed (Participants) | 19 | 17
minutes
  First Night | 193.42 (55.529) | 198.41 (43.364)
  Second Night | 214.89 (56.916) | 188.88 (45.862)

10. Secondary Outcome: Stage N3 (Min)
Description: Stage N3 is considered as 'deep sleep'. It is sometimes referred as slow wave sleep.
Time Frame: per night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FRESCA Mask First Night | CPAP Second Night | CPAP Mask First Night | FRESCA Mask Second Night
Number analyzed (Participants) | 19 | 17
minutes
  First Night | 59.21 (44.065) | 60.35 (50.447)
  Second Night | 56.21 (48.433) | 42.94 (39.366)

11. Secondary Outcome: REM (Min)
Description: The exact function of the REM is uncertain. However, it occupies approximately 25% of the total sleep time. REM sleep cycles occur every 90 to 120 min throughout the night with progressively increasing periods of time. REM sleep is associated with more frequent and longer duration apneas, hypopneas, and severe hypoxemia
Time Frame: per night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FRESCA Mask First Night | CPAP Second Night | CPAP Mask First Night | FRESCA Mask Second Night
Number analyzed (Participants) | 19 | 17
minutes
  First Night | 60.63 (23.150) | 72.29 (26.343)
  Second Night | 93.79 (31.101) | 58.82 (25.914)

ADVERSE EVENTS:
Time Frame: All adverse events were record from the time they occurred.
Description: The 47 participants at risk include the 36 who completed the two sleep nights and the 11 who withdrew early.
Groups:
- FRESCA Mask: Each patient used both devices, the analysis of the Adverse Events is recorded for both technology. This arm is associated with the FRESCA Mask.
- CPAP Mask: Each patient used both devices, the analysis of the Adverse Events is recorded for both technology. This arm is associated with the CPAP Mask.
Arm/Group | FRESCA Mask | CPAP Mask
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 4/47 | 0/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FRESCA Mask (N=47) | CPAP Mask (N=47)
Difficulty breathing through study device (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No